CLINICAL TRIAL: NCT03166501
Title: NMDA Receptor Modulation for Hyperarousal in PTSD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sanjay Johan Mathew, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36371; 1R61MH110540-01 (NIH)
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2019-11

CONDITIONS: Depression; Post Traumatic Stress Disorder
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic | interventions — AZD6765

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Lanicemine 100mg Intravenous
  Interventions: Drug: Lanicemine
- Placebo (Placebo Comparator): Normal saline Intravenous
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lanicemine — Three 60 min parenteral infusions over a 5 day period
  Other Names: BHV-5500
  Arms: Treatment
Drug: Placebo — Three 60 min parenteral infusions over a 5 day period
  Other Names: Baxter
  Arms: Placebo

SUMMARY:
This Phase 1b study examines the safety and efficacy of parenterally-administered lanicemine in a parallel-arm, randomized, double-blind, placebo-controlled trial in adult patients (N=24) with significant PTSD symptoms and elevated anxiety potentiated startle (APS). Investigator hypothesize that lanicemine (100 mg) displays a normalization of APS following three infusions over 5 non-consecutive days. If target engagement is demonstrated and the drug is safe and tolerable in this patient population, investigator will proceed to a larger POC study.

DETAILED DESCRIPTION:
This study aims to provide a rigorous test of functional target engagement and "go/no go" milestones for a subsequent POC trial. Investigator will conduct a parallel-arm, randomized, double-blind, placebo-controlled study to assess lanicemine (100 mg) with respect to a functional pharmacodynamic readout of target engagement (APS). Twenty-four patients with significant PTSD symptoms and elevated APS will be randomized to one of 2 treatment groups [placebo or 100 mg], and undergo three 60 min parenteral infusions over a 5 day period. APS and other neurophysiological biomarkers will be tested before and after the 1st and 3rd treatment.

Primary Objective is to examine, relative to placebo, whether lanicemine will demonstrate normalization of the APS response following three treatments.

Secondary Objectives are to examine, relative to placebo, whether lanicemine will demonstrate effects on P50 auditory evoked potentials, gamma band EEG, and Mismatch Negativity. Investigator also explore whether target engagement will mediate the effect of treatment on CAPS-5 scores.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Patients must provide acceptable proof of identity documentation to confirm initials and date of birth
3. Male and female patients aged 21 to 65 years, inclusive.
4. All male patients who are sexually active must agree to use a double barrier method of contraception (condom with spermicide) from the first dose of IP until 12 weeks after their last dose. All females must have a negative serum pregnancy test. Women of childbearing potential (WOCBP, see below) must use a highly effective form of birth control plus the use of a condom by the male sexual partner, reviewed and approved by the PI. The highly effective form of birth control includes: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective IUD/IUS, Depo-Provera injections, oral contraceptive, and Evra Patch or Nuvaring. Women should be on a stable method of birth control for a minimum of 3 months , prior to randomization and 3 months after the last dose of IP.

   Women of non-childbearing potential. Women of non-childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they are amenorrheic for 12 months prior to randomization without an alternative medical cause. The following age-specific requirements apply:

   Women < 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.

   Women ≥ 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
5. CAPS-5 score ≥ 25 and CGI-S ≥ 4 at Screening and Randomization
6. Anxiety Potentiated Startle T-score ≥ 2.8.
7. Psychotropic medications must remain at a stable dose for at least 42 days prior to screening, without clinically significant adjustment.
8. Be able to understand and comply with the requirements of the study, as judged by the investigator

Exclusion Criteria:

1. Patients who are currently participating in another clinical study in which the patient is exposed to an investigational or non-investigational drug or device, or have done so within the last 30 days prior to screening.
2. Patients who have no regular contact with an adult who could come to the patient's aid should an urgent need arise.
3. Patients with a history of DSM-5 diagnosis of bipolar disorder, schizophrenia or schizoaffective disorder, or currently exhibiting psychotic symptoms associated with depression; dementia or suspicion thereof, is also exclusionary.
4. Currently being treated with MAOIs, lithium, divalproex, carbamazepine, barbiturates, or benzodiazepines. Patients taking medications with known activity at the NMDA or AMPA glutamate receptor [eg, riluzole, amantadine, lamotrigine, memantine, topiramate, dextromethorphan, D-cycloserine], or the mu-opioid receptor.
5. Patients who meet DSM-5 criteria for substance use disorder (amphetamines, cocaine, hallucinogens, inhalants, opioids, sedatives/hypnotics/anxiolytics) within 1 month prior to screening. Patients with a positive urine drug screen (UDS) are excluded except for patients testing positive for prescribed medications that are otherwise permitted and there is no evidence of misuse or abuse. Patients can be re-tested only if either the initial opiate or barbiturate result is positive and they have a prescription, but the patient should be excluded if the result is still positive at the second test. Patients with positive UDS for drug(s) legally available by prescription must provide evidence of prescription for the drug(s).
6. Patients with a binge-pattern of alcohol use which makes them at risk for withdrawal-related seizures. Also, significant alcohol withdrawal symptoms that require medical detoxification.
7. Patients with a suicide attempt within the last 3 months or at imminent risk of suicide and not suitable for an outpatient study, in the judgment of the investigator.
8. Patients who are pregnant or lactating.
9. Clinically significant laboratory value, physical examination, or ECG that signifies a major medical illness that is unstable or inadequately controlled, or that may put the subject at risk during the study in the judgment of the investigator. Hypothyroidism is permitted if corrected and the patient is on a stable treatment regimen for a minimum of 6 months.
10. Systolic BP < 85 or > 160 mmHg or diastolic BP > 100 mmHg or heart rate < 50 or >105 beats per minute at Screening or Randomization. Exclusionary values may be repeated once.
11. QTcF (Fridericia-corrected) ≥ 450 msec at Screening or Randomization. Exclusionary values may be repeated once.
12. Patients with any history of seizure disorder (except for febrile seizures in childhood) or traumatic brain injury.
13. Previous exposure to lanicemine.
14. Patients with a personality disorder which in the opinion of the investigator has a major impact on the patient's current psychiatric status and would preclude safe study participation.
15. Body mass index (BMI) ≥ 40 kg/m2

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Primary Objective | 24 months
  Primary Objective is to examine, relative to placebo, whether lanicemine will demonstrate normalization of the APS response following three treatments.

SECONDARY OUTCOMES:
Secondary Objectives (1/4) | 24 months
  To examine, relative to placebo, whether lanicemine will demonstrate effects on P50 auditory evoked potentials
Secondary Objectives (2/4) | 24 months
  To examine, relative to placebo, whether lanicemine will demonstrate effects on gamma band EEG
Secondary Objectives (3/3) | 24 months
  To examine, relative to placebo, whether lanicemine will demonstrate effects on Mismatch Negativity
Secondary Objectives (4/4) | 24 months
  Also explore whether target engagement will mediate the effect of treatment on CAPS-5 scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873
- [Derived] Ramakrishnan N, Lijffijt M, Green CE, Balderston NL, Murphy N, Grillon C, Iqbal T, Vo-Le B, O'Brien B, Murrough JW, Swann AC, Mathew SJ. Neurophysiological and clinical effects of the NMDA receptor antagonist lanicemine (BHV-5500) in PTSD: A randomized, double-blind, placebo-controlled trial. Depress Anxiety. 2021 Nov;38(11):1108-1119. doi: 10.1002/da.23194. Epub 2021 Jul 12. PMID 34254405
- [Derived] Murphy N, Lijffijt M, Ramakrishnan N, Vo-Le B, Vo-Le B, Iqbal S, Iqbal T, O'Brien B, Smith MA, Swann AC, Mathew SJ. Does mismatch negativity have utility for NMDA receptor drug development in depression? Braz J Psychiatry. 2022 Jan-Feb;44(1):61-73. doi: 10.1590/1516-4446-2020-1685. PMID 33825765
- [Derived] Lijffijt M, Green CE, Balderston N, Iqbal T, Atkinson M, Vo-Le B, Vo-Le B, O'Brien B, Grillon C, Swann AC, Mathew SJ. A Proof-of-Mechanism Study to Test Effects of the NMDA Receptor Antagonist Lanicemine on Behavioral Sensitization in Individuals With Symptoms of PTSD. Front Psychiatry. 2019 Dec 13;10:846. doi: 10.3389/fpsyt.2019.00846. eCollection 2019. PMID 31920733